CLINICAL TRIAL: NCT03553602
Title: A Phase I/II Study of Salvage High-dose-rate Brachytherapy, ExternAl Beam COmbined and Short-term Hormonal Therapy for the Treatment of Node-positive Locally Recurrent Prostate Cancer After Prior Definitive Radiotherapy
Brief Title: HDR Brachytherapy, EBRT and STAD for the Treatment of Prostate Cancer
Acronym: BEACON
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was stopped for feasibility
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Abhishek A. Solanki, Assistant Professor, Loyola University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 210546
Record Dates: First submitted 2018-05-30; First posted 2018-06-12 (Actual); Results first posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer - Recurrent
Keywords: Prostate Cancer; HDR brachytherapy; Recurrent Prostate Cancer; Oligometastasis; Salvage Brachytherapy; Salvage Radiotherapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- HDR Brachytherapy + EBRT + STAD (Experimental): Day 1: HDR Brachytherapy implant: 2 fractions of 12 Gy to prostate/ proximal SV.
  EBRT: 50.4 Gy in 28 fractions to the pelvic lymph nodes +/- para-aortic nodes, with SIB up to 70 Gy to the PET positive lesions.
  6 months hormonal therapy(LHRH agonist and antiandrogen [until the end of radiotherapy])
  Interventions: Drug: HDR Brachytherapy + EBRT + STAD

INTERVENTIONS:
Drug: HDR Brachytherapy + EBRT + STAD — HDR Brachytherapy implant: 2 fractions of 12 Gy to the prostate/ proximal SV.
  EBRT: 50.4 Gy in 28 fractions to the pelvic lymph nodes +/- para-aortic nodes, with SIB up to 70 Gy to the PET- positive lesions.
  6 months hormonal therapy(LHRH agonist and anti-androgen[until end of radiotherapy])

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of combining high-dose-rate (HDR) brachytherapy with external beam radiotherapy (EBRT) to the pelvis and 6 months of hormonal therapy, otherwise known as short term androgen deprivation therapy (STAD), as treatment for prostate cancer that has come back in the prostate and pelvic lymph nodes after prior radiotherapy. The study will examine the side effects of the treatment as well as the ability of the treatment to get rid of the cancer. This involves the placement of a radioactive material in the affected area of the prostate temporarily, and then is subsequently removed using a minimally invasive technique. Participants will also receive external radiation for 5 weeks targeting the pelvis and giving a higher dose each day to the suspicious lymph nodes on PET scan. Radiation therapy will start approximately 2 months after the start of the Androgen Deprivation Therapy (hormone therapy). The hormone therapy consists of two medications, an oral medication taken daily 2 months before starting radiation therapy until the last of the radiation therapy and an injection of a medication which is given 2 months prior to the start of radiation. Patient are then followed at specific time intervals to evaluate the treatment side effects and cancer control

DETAILED DESCRIPTION:
Salvage regional and local radiation is frequently utilized across multiple disease sites in oncology for patients who have failed initial radiotherapy. However, in prostate cancer, due to the concern that nodal involvement is a manifestation of widespread distant disease, this type of approach has not typically been pursued. However, with newer imaging modalities such as fluciclovine PET, PSMA pet, and C11 PET, physicians are identifying nodal disease and excluding distant disease better than they ever have before. Thus, in the modern era regional control may translate to improved long-term biochemical control, and prevent the morbidity and mortality associated with clinical progression of recurrent prostate cancer

Thus, in patients who recur both in the prostate and in the pelvic lymph nodes, treating both with radiation could result in meaningful clinical efficacy for patients-similar to other disease sites. However, there are limited data exploring the feasibility and safety of this combination. Therefore, the investigators are conducting this trial, which combines salvage HDR brachytherapy to the local recurrence of the prostate cancer with EBRT to the pelvic lymph nodes, and short-term hormonal therapy, in this group of patients. The investigators hypothesize that this approach can safely be performed without excess toxicity.

Once a patient is deemed eligible for the study and has signed the informed consent form, the patient will start hormone therapy with a LHRH Agonist medication which is an intramuscular injection which patients will receive every 3-6 months for 6 months. Within 10 days of the LHRH injection the patient must start an anti-androgen pill and will take the pill once a day until the last day of radiation. Radiation Therapy will start approximate 2 months after the start of the hormone therapy. Patients will undergo 2 implants with 1 fraction of 12 Gy delivered with each implant, scheduled 1-2 weeks apart when possible, although longer or shorter intervals are acceptable with PI approval. The implant procedure will be done under general anesthesia. Patients will also receive the external beam radiotherapy (for 5 weeks), starting before or after the brachytherapy treatment. Patients will also be asked to complete 2 short quality of life questionnaires before they receive treatment and at follow up visits. Patient will follow up with the radiation oncologist for an exam at 1 month, 3 months, 6 months and 12 months after treatment and then every 6 months for 4 more years then annually thereafter.

ELIGIBILITY:
Inclusion Criteria

* Biopsy proven locally recurrent adenocarcinoma of the prostate after the completion of definitive radiation therapy for initially diagnosed prostate cancer.
* Initial cancer diagnosis that fits these specific criteria:

  * Stages cT1-T3a
  * Nx or N0
  * Mx or M0
* Eligible initial definitive radiotherapy modalities include:

  * External beam radiotherapy, with photon or proton beam therapy
  * Definitive Brachytherapy
  * Stereotactic Body Radiotherapy
* Fluciclovine-positive pelvic nodes (as determined by an interpreting radiologist or nuclear medicine physician) in the pelvic nodal region (defined as the pelvic nodal regions up to the common iliac nodal region) without any evidence of lymph node involvement outside of this area or distant metastases
* Candidate for hormonal therapy.
* Current ECOG Performance status Scale 0-2 (Appendix D)
* Current International Prostate Symptom Score (IPSS) < 20 (Appendix B)
* Age >18
* The patient must be medically suitable to receive general or spinal anesthesia.
* AST, ALT, and alkaline phosphatase < 2 x upper institutional limit within 3 months of registration.
* The patient must be able and willing to sign a study-specific written informed consent form before study entry.

Exclusion Criteria

* Preregistration radiation-related GI or GU toxicity (for any reason) grade ≥ 3 as defined in CTCAE version 4.03. That is, grade ≥ 3 GU or GI toxicity after first course of radiotherapy
* Treatment to a "whole pelvis" field with initial radiotherapy
* Patients with distant metastases (such as to the bone, visceral organs, and lymph nodes other than the pelvic nodes including the common iliac nodes).
* Patients receiving any other investigational agents.
* Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, severely symptomatic congestive heart failure, cardiac arrhythmia, recent myocardial infarction in last 6 months, or psychiatric illness/social situations that could limit compliance with study requirements.
* Patients who have received chemotherapy or immunotherapy within one month prior to study enrollment, other than ADT.

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2024-07-26 (Actual); Study Completion 2024-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abhishek Solanki, MD, Principal Investigator — Loyola University Chicago
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peduzzi P, Concato J, Kemper E, Holford TR, Feinstein AR. A simulation study of the number of events per variable in logistic regression analysis. J Clin Epidemiol. 1996 Dec;49(12):1373-9. doi: 10.1016/s0895-4356(96)00236-3. PMID 8970487
- [Background] Simon R. Optimal two-stage designs for phase II clinical trials. Control Clin Trials. 1989 Mar;10(1):1-10. doi: 10.1016/0197-2456(89)90015-9. PMID 2702835
- [Background] Savir-Baruch B, Zanoni L, Schuster DM. Imaging of Prostate Cancer Using Fluciclovine. PET Clin. 2017 Apr;12(2):145-157. doi: 10.1016/j.cpet.2016.11.005. Epub 2017 Jan 23. PMID 28267449
- [Background] Suardi N, Gandaglia G, Gallina A, Di Trapani E, Scattoni V, Vizziello D, Cucchiara V, Bertini R, Colombo R, Picchio M, Giovacchini G, Montorsi F, Briganti A. Long-term outcomes of salvage lymph node dissection for clinically recurrent prostate cancer: results of a single-institution series with a minimum follow-up of 5 years. Eur Urol. 2015 Feb;67(2):299-309. doi: 10.1016/j.eururo.2014.02.011. Epub 2014 Feb 18. PMID 24571959
- [Background] Lin D, Wei L, Ying Z. Checking the Cox Model with Cumulative Sums of Martingale-Based Residuals. Biometrika. 1993;80:557-572.
- [Background] Rigatti P, Suardi N, Briganti A, Da Pozzo LF, Tutolo M, Villa L, Gallina A, Capitanio U, Abdollah F, Scattoni V, Colombo R, Freschi M, Picchio M, Messa C, Guazzoni G, Montorsi F. Pelvic/retroperitoneal salvage lymph node dissection for patients treated with radical prostatectomy with biochemical recurrence and nodal recurrence detected by [11C]choline positron emission tomography/computed tomography. Eur Urol. 2011 Nov;60(5):935-43. doi: 10.1016/j.eururo.2011.07.060. Epub 2011 Aug 3. PMID 21840116
- [Background] Chen CP, Weinberg V, Shinohara K, Roach M 3rd, Nash M, Gottschalk A, Chang AJ, Hsu IC. Salvage HDR brachytherapy for recurrent prostate cancer after previous definitive radiation therapy: 5-year outcomes. Int J Radiat Oncol Biol Phys. 2013 Jun 1;86(2):324-9. doi: 10.1016/j.ijrobp.2013.01.027. Epub 2013 Mar 6. PMID 23474112
- [Background] Yamada Y, Kollmeier MA, Pei X, Kan CC, Cohen GN, Donat SM, Cox BW, Zelefsky MJ. A Phase II study of salvage high-dose-rate brachytherapy for the treatment of locally recurrent prostate cancer after definitive external beam radiotherapy. Brachytherapy. 2014 Mar-Apr;13(2):111-6. doi: 10.1016/j.brachy.2013.11.005. Epub 2013 Dec 25. PMID 24373762
- [Background] Crook J, Pisansky TM, Clinic M, et al. Nrg Oncology Rtog 0526.; 1818.
- [Background] Beyer DC. Permanent brachytherapy as salvage treatment for recurrent prostate cancer. Urology. 1999 Nov;54(5):880-3. doi: 10.1016/s0090-4295(99)00241-1. PMID 10565751
- [Background] Grado GL, Collins JM, Kriegshauser JS, Balch CS, Grado MM, Swanson GP, Larson TR, Wilkes MM, Navickis RJ. Salvage brachytherapy for localized prostate cancer after radiotherapy failure. Urology. 1999 Jan;53(1):2-10. doi: 10.1016/s0090-4295(98)00492-0. PMID 9886580
- [Background] Parekh A, Graham PL, Nguyen PL. Cancer control and complications of salvage local therapy after failure of radiotherapy for prostate cancer: a systematic review. Semin Radiat Oncol. 2013 Jul;23(3):222-34. doi: 10.1016/j.semradonc.2013.01.006. PMID 23763889
- [Background] Michalski JM, Pisansky TM, Lawton CAF, Potters L. Prostate Cancer. Clin Radiat Oncol. 2016:1038-1095.e18. doi:10.1016/B978-0-323-24098-7.00053-8.
- [Background] Wirth MP, Hakenberg OW, Froehner M. Antiandrogens in the treatment of prostate cancer. Eur Urol. 2007 Feb;51(2):306-13; discussion 314. doi: 10.1016/j.eururo.2006.08.043. Epub 2006 Sep 11. PMID 17007995
- [Background] Ahmadi H, Daneshmand S. Androgen deprivation therapy for prostate cancer: long-term safety and patient outcomes. Patient Relat Outcome Meas. 2014 Jul 5;5:63-70. doi: 10.2147/PROM.S52788. eCollection 2014. PMID 25045284
- [Background] Zumsteg ZS, Spratt DE, Romesser PB, Pei X, Zhang Z, Kollmeier M, McBride S, Yamada Y, Zelefsky MJ. Anatomical Patterns of Recurrence Following Biochemical Relapse in the Dose Escalation Era of External Beam Radiotherapy for Prostate Cancer. J Urol. 2015 Dec;194(6):1624-30. doi: 10.1016/j.juro.2015.06.100. Epub 2015 Jul 10. PMID 26165583
- [Background] Zelefsky MJ, Kuban DA, Levy LB, Potters L, Beyer DC, Blasko JC, Moran BJ, Ciezki JP, Zietman AL, Pisansky TM, Elshaikh M, Horwitz EM. Multi-institutional analysis of long-term outcome for stages T1-T2 prostate cancer treated with permanent seed implantation. Int J Radiat Oncol Biol Phys. 2007 Feb 1;67(2):327-33. doi: 10.1016/j.ijrobp.2006.08.056. Epub 2006 Nov 2. PMID 17084558
- [Background] Shipley WU, Thames HD, Sandler HM, Hanks GE, Zietman AL, Perez CA, Kuban DA, Hancock SL, Smith CD. Radiation therapy for clinically localized prostate cancer: a multi-institutional pooled analysis. JAMA. 1999 May 5;281(17):1598-604. doi: 10.1001/jama.281.17.1598. PMID 10235152
- [Background] Demanes DJ, Martinez AA, Ghilezan M, Hill DR, Schour L, Brandt D, Gustafson G. High-dose-rate monotherapy: safe and effective brachytherapy for patients with localized prostate cancer. Int J Radiat Oncol Biol Phys. 2011 Dec 1;81(5):1286-92. doi: 10.1016/j.ijrobp.2010.10.015. Epub 2011 Feb 9. PMID 21310546
- [Background] Henriquez I, Sancho G, Hervas A, Guix B, Pera J, Gutierrez C, Abuchaibe O, Martinez-Monge R, Tormo A, Polo A. Salvage brachytherapy in prostate local recurrence after radiation therapy: predicting factors for control and toxicity. Radiat Oncol. 2014 Apr 30;9:102. doi: 10.1186/1748-717X-9-102. PMID 24885287
- [Background] Tward JD, Kokeny KE, Shrieve DC. Radiation therapy for clinically node-positive prostate adenocarcinoma is correlated with improved overall and prostate cancer-specific survival. Pract Radiat Oncol. 2013 Jul-Sep;3(3):234-240. doi: 10.1016/j.prro.2012.11.011. Epub 2013 Jan 28. PMID 24674370
- [Background] Meng MB, Wang HH, Zaorsky NG, Zhao XZ, Wu ZQ, Jiang B, Song YC, Zhuang HQ, Li FT, Zhao LJ, Wang CL, Li K, Wang P, Yuan ZY. Clinical evaluation of stereotactic radiation therapy for recurrent or second primary mediastinal lymph node metastases originating from non-small cell lung cancer. Oncotarget. 2015 Jun 20;6(17):15690-703. doi: 10.18632/oncotarget.3704. PMID 25881546
- [Background] Parks J, Kloecker G, Woo S, Dunlap NE. Stereotactic Body Radiation Therapy as Salvage for Intrathoracic Recurrence in Patients With Previously Irradiated Locally Advanced Non-Small Cell Lung Cancer. Am J Clin Oncol. 2016 Apr;39(2):147-53. doi: 10.1097/COC.0000000000000039. PMID 24457534
- [Background] Hearn JW, Videtic GM, Djemil T, Stephans KL. Salvage stereotactic body radiation therapy (SBRT) for local failure after primary lung SBRT. Int J Radiat Oncol Biol Phys. 2014 Oct 1;90(2):402-6. doi: 10.1016/j.ijrobp.2014.05.048. Epub 2014 Jul 10. PMID 25017480
- [Background] Prostate Cancer Statistics. 2016.

RESULTS

PARTICIPANT FLOW:
Groups:
- HDR Brachytherapy + EBRT + STAD: Day 1: HDR Brachytherapy implant: 2 fractions of 12 Gy to prostate/ proximal SV.
  EBRT: 50.4 Gy in 28 fractions to the pelvic lymph nodes +/- para-aortic nodes, with SIB up to 70 Gy to the PET positive lesions.
  6 months hormonal therapy(LHRH agonist and antiandrogen [until the end of radiotherapy])
  HDR Brachytherapy + EBRT + STAD: HDR Brachytherapy implant: 2 fractions of 12 Gy to the prostate/ proximal SV.
  EBRT: 50.4 Gy in 28 fractions to the pelvic lymph nodes +/- para-aortic nodes, with SIB up to 70 Gy to the PET- positive lesions.
  6 months hormonal therapy(LHRH agonist and anti-androgen[until end of radiotherapy])
Period: Overall Study
Arm/Group | HDR Brachytherapy + EBRT + STAD
Started | 3
Completed | 2
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | HDR Brachytherapy + EBRT + STAD
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Genitourinary Toxicity
Description: The primary outcome in this study is the number of participants with an acute grade ≥3 radiation-related genitourinary toxicity as described by the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
Time Frame: 24 months
Population: Two participants completed the month 24 assessment
Measure: Count of Participants; unit: Participants
Arm/Group | HDR Brachytherapy + EBRT + STAD
Number analyzed (Participants) | 2
Participants | 0

2. Secondary Outcome: Gastrointestinal Toxicity
Description: A secondary outcome in this study is the number of participants with an acute grade ≥3 radiation-related gastrointestinal toxicity as described by the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
Time Frame: 24 months
Population: Two participants completed the month 24 assessment
Measure: Count of Participants; unit: Participants
Arm/Group | HDR Brachytherapy + EBRT + STAD
Number analyzed (Participants) | 2
Participants | 1

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 4 years
Arm/Group | HDR Brachytherapy + EBRT + STAD
All-Cause Mortality (participants affected / at risk) | 1/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-10-23): https://cdn.clinicaltrials.gov/large-docs/02/NCT03553602/Prot_SAP_002.pdf
  • Informed Consent Form (2023-11-15): https://cdn.clinicaltrials.gov/large-docs/02/NCT03553602/ICF_003.pdf